CLINICAL TRIAL: NCT01795313
Title: Immunotherapy for Recurrent Ependymomas in Children Using Human Leukocyte Antigen (HLA)-A2 Restricted Tumor Antigen Peptides in Combination With Imiquimod
Brief Title: Immunotherapy for Recurrent Ependymomas in Children Using Tumor Antigen Peptides With Imiquimod
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed supratentorial arm prematurely secondary to lack of enrollment
Sponsor: James Felker (Other)
Collaborators: Solving Kids' Cancer (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, James Felker, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100001; R01CA174858 (NIH); PRO12050422 (Other: Former IRB protocol ID)
Record Dates: First submitted 2013-02-12; First posted 2013-02-20 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ependymoma
MeSH Terms: conditions — Ependymoma | interventions — Imiquimod; Enzyme-Linked Immunosorbent Assay; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Intervention Model Description: This is a pilot study to assess tolerability of our vaccine regimen in children with ependymomas initially arising above or below the tentorium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLA-A2 restricted tumor antigen vaccine (Experimental): This is a single-arm study of a HLA-A2 restricted tumor antigen peptide vaccine, administered in conjunction with imiquimod
  Interventions: Biological: HLA-A2 restricted synthetic tumor antigen; Drug: Imiquimod; Other: enzyme-linked immunosorbent assay; Other: flow cytometry; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: HLA-A2 restricted synthetic tumor antigen
Drug: Imiquimod
Other: enzyme-linked immunosorbent assay
Other: flow cytometry
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
The purpose of this study is to see if vaccination with HLA-A2 restricted peptides, combined with the immunoadjuvant imiquimod is safe and can induce immune responses in children with recurrent ependymomas. Eligible patients are stratiﬁed by primary tumor location.

ELIGIBILITY:
Inclusion Criteria: All grades of ependymoma are eligible.

* Patients must have recurrent/progressive ependymoma that has progressed or recurred after initial adjuvant therapy.
* HLA-A2 positive based on flow cytometry performed at the University of Pittsburgh.
* Patients must have previously received standard initial therapy including attempted gross total resection, where safely feasible, and in appropriate circumstances (e.g., those older than one year at initial diagnosis, with non-metastatic tumors and at least microscopic residual disease), involved field fractionated radiation therapy (RT). Patients may have received re-irradiation but not to the index lesion within 4 weeks.
* Patients must be clinically stable and off or on low-dose (no more than 0.1 mg/kg/day, max 4 mg/day Dexamethasone) corticosteroid for at least one week prior to study registration.
* Patients must be ≥ 12 months and <22 years of age at the time of study registration.
* Patients must have a performance status of ≥ 70; (Karnofsky if > 16 years and Lansky if ≤ 16 years of age).
* Patients may have non-bulky, asymptomatic metastatic disease.
* Males and females must agree to use effective birth control methods during the course of vaccination (from the first vaccine to two weeks after the last vaccine).
* Patients must be free of systemic infection requiring IV antibiotics at the time of registration and off IV antibiotics for at least 7 days prior to registration.
* Patients must have adequate organ function as measured by:

  * Bone marrow: Absolute neutrophil count (ANC) > 1,000/µl; Platelets > 100,000/µl (transfusion independent); Absolute lymphocyte count (ALC) ≥ 500/µl; Hemoglobin >8 g/dl (may be transfused).
  * Hepatic: bilirubin ≤ 1.5x institutional normal for age; serum glutamate pyruvate transaminase (SGPT) < 3x institutional normal
  * Renal: Serum creatinine based on age or creatinine clearance or radioisotope glomerular filtration rate (GFR) > 70 ml/min/1.73 m²
* Patients must have recovered from the toxic effects of prior therapy and be at least 3 weeks from the last dose of standard cytotoxic chemotherapy or myelosuppressive biological therapy, at least one week from the last dose of non-myelosuppressive biological therapy and at least 4 weeks from the completion of radiation therapy.
* Patients must have no overt cardiac, gastrointestinal, pulmonary, or psychiatric disease.

Patients must be willing to travel to Pittsburgh to receive the vaccine. Visits: Every 3 weeks x 9, then every 6 weeks x 12 depending on response/side effects

Exclusion Criteria:

* Patients living outside of North America are not eligible.
* Patients must be off concurrent treatment or medications for at least 1 week including: Interferon (e.g. Intron-A®), allergy desensitization injections, growth factors (e.g. Procrit®, Aranesp®, Neulasta®), interleukins (e.g. Proleukin®), and any investigational therapeutic medication.
* Patients must not have a history of any immune system disorder or laboratory abnormality or any condition that could potentially alter immune function.
* Use of immunosuppressives within four weeks prior to study entry or anticipated use of immunosuppressive agents. Patients must be on no more than 0.1 mg/kg/day, max 4 mg/day dexamethasone for at least one week before study registration. Topical corticosteroids are acceptable.
* Patients with a known immune deficiency.
* Pregnancy or breastfeeding. Female patients who are post-menarchal must have a documented negative pregnancy test.
* Tetanus vaccine during therapy or within 1 week prior to enrollment.
* Patients who have received prior immunotherapy.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with unacceptable toxicity | 2 years
  Grade 3 or 4 non-hematological toxicities.

SECONDARY OUTCOMES:
Tumor-associated antigen-specific T-cell | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Felker, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States